CLINICAL TRIAL: NCT06970691
Title: is Generalized Aggressive Periodontitis an Endless Disease When Does it Stop
Status: Completed | Type: Observational
Sponsor: Rasha Wagih (Other)
Responsible Party: Sponsor-Investigator, Rasha Wagih, Head of periodontology department, Badr University
Organization: Badr University (Other)
Other Study IDs: 240418-89
Record Dates: First submitted 2025-03-17; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Aggressive Periodontitis, Generalized
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: panoramic radiograph — Panoramic radiographs for aggressive periodontitis previously diagnosed cases were interpreted by single examiner (NY). The included radiographs had to fulfill the following; 1) sufficient image quality; 2) All teeth with the surrounding alveolar bone had to be clear enough to facilitate alveolar bone tracing; 3) Only pre-operative radiographs were enrolled (before the surgical management of bony defects).

SUMMARY:
Background: Inquiring thoroughly and systematically for evidence supporting the mechanism, time span, onset, or ending events of generalized aggressive periodontitis. The aim of the current retrospective cross-sectional study was to set temporal boundaries of the generalized form of aggressive periodontitis based on eruption time of permanent teeth via panoramic radiographs.

Methods: based on the Egyptian chronology, the primary outcome of the current retrospective study was to assess the correlation between the eruption sequence and the temporal borders of the disease as well as the prevalence of destructive events in accordance to the eruption schedule. The first affected tooth, the last affected tooth, the first unaffected tooth, the number of affected teeth, the presence of interrupted tooth all are factors that extracted from the panoramic radiographs.

DETAILED DESCRIPTION:
During the last decades, progressive lines of thinking were proposed by generations of brilliant periodontists who tried to describe the aggressive destruction of periodontal tissues. Periodontitis was basically described 2000 years ago but in 18th century, signs and symptoms of periodontitis were firstly recorded.

History of aggressive periodontitis At the beginning of 19th century, alveolar pyorrhea was a term created and explained by two different schools; the European school has described it as a disease which is not affected by local factors while the American school has described local factors especially salivary calculus as the main cause behind alveolar pyorrhea.

Later by the development of histological, radio graphical and microbiological analysis, three other explanation were raised; school of atrophy and degeneration, school of occlusal trauma and school of infection. The European School has supported the theory of atrophy and degeneration especially in young individuals. Their explanation was mainly based on the histological studies which concluded that alveolar bone loss is the primary crucial point in periodontal disease preceded by gingival ulceration and inflammation. Pocket formation and epithelial proliferation are secondary events. Furthermore, they also reported that inflammation and suppuration are strongly connected to the presence of external irritation and entitled it ''Diffuse atrophy''.

Classification of Aggressive periodontitis In 80s and 90s, numerous classifications with various staging and subtypes had been conducted which were not based upon the true diagnostic background. In 1986, the American academy of periodontology acknowledged the exclusion of rapidly progressive periodontitis and added prepubertal periodontitis as a subclass to juvenile periodontitis. In 1989, the American academy classification was modified. They proposed early onset periodontitis to include both prepubertal, juvenile and rapidly progressive periodontitis and added periodontitis associated with systemic disease as separate entity. In 1989, Topic subdivided the periodontal conditions into acute and chronic. The acute condition included periodontal abscess, pericoronitis while the chronic condition included periodontitis (simplex, complex and generalized forms), localized forms (juvenile, post-juvenile and prepubertal) and symptomatic. The latter classification was lacking essential details concerning the periodontal diseases. In 1994, the European Workshop on Periodontology condensed the previous classes into; early onset, adult and necrotizing periodontitis. In 1997, the Committee of American Academy of Periodontology had set a plan to revise the previously proposed classifications.

Sub-typing of aggressive periodontitis Early onset description of periodontitis was mainly based on the influence of patient's age at the time of reporting the evolution of symptoms added to the short-term period in which uppermost destructive events had happened. In 1989 classification, early onset periodontitis was sub-categorized as pre-pubertal juvenile and rapidly progressive periodontitis. Both sub-categories approved to be either localized or generalized.

In 1999, Armittage classification replaced the term ''Early onset periodontitis, EOP'' with ''Aggressive periodontitis''. The term Aggressive periodontitis described the early onset events that cause severe and rapid periodontal damage in young patients. Aggressive periodontitis was directly classified into localized; LJP (classical incisor-molar pattern) and generalized forms. Here, the ages as well as the time scale period of destruction were not determinant factors for the nature of the disease as in 1989 classification. It was mainly based on the degree and distribution of destruction. No difference was defined to differentiate primary or permanent teeth affection.

In 2018, the latest classification added the molar-incisor pattern (MIPP) as a separate subtype of severe periodontitis from the localized form. It affects only the incisors and molars.

Difference between Chronic and aggressive periodontitis According to 1999 classification, there were four main features that categorized aggressive over the chronic one. Firstly, the onset; where aggressive periodontitis begins its manifestation in a relatively young age. Secondly, the rate of destruction is more rapid in aggressive form. Thirdly, the familial background in aggressive is more prone to affect more than one person in the same family. Fine et al., 2018, in their latest classification, combined both diseases into only one category called ''Periodontitis'' and added a staging and grading system. The authors could not stand totally against the existence of aggressive periodontitis nature as a separate unique entity with the explicit, lesions' location, familial background, rate of progression, age of onset and the deposits amount. The combination of the 2 categories was explained due to the absence of enough solid evidence for aggressive periodontitis describing it as a separate entity.

Unfortunately, from the knowledge in the literature, aggressive periodontitis, as a disease, represents a gap of knowledge. The nature of the disease, the incidence of initiation, when it ends, if it is accompanied by other medical problems, and if it is a solitary manifestation of a rare independent disease that is not related to any other body organs, all are questions that couldn't find a clue.

Research hypothesis In the current research, we propose that generalized aggressive periodontitis, begins at or before the eruption of the first permanent tooth. Then, it continues without quiescence period (not interrupted) till it stops exactly when the immune system shows enough maturation. We speculated that the eruption time scale of the affected tooth translates disease activity during this period while eruption of unaffected permanent tooth indicates point time of disease suppression.

ELIGIBILITY:
Inclusion Criteria:

* patients with generalized ggressive perioodntitis only
* Panoramic view is a must
* Patient age ≥ 18 years
* both genders were enrolled
* Radiographic evidence of bony defects was compulsory for inclusion.

Exclusion Criteria:

* patients who did not have panoramic radiograph in their files
* Patients less than 18 years are not included

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All radiographic panoramic records of patients, who were previously clinically diagnosed as generalized aggressive periodontitis, were included. Fills with other radiographic records other than panoramic views were excluded. For this study, the enrolled patients' age was selected ≥ 18 years of both genders. Radiographic evidence of bony defects was compulsory for inclusion.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
the radiographic eruption date of the first and the last affected teeth | 4 years
  based on panoramic view of each patient, the radiographic eruption date of the mentioned teeth was determined.

SECONDARY OUTCOMES:
The radiographic status of the supporting structures of third molars | 4 years
  based on the panormaic view of each patient, the condiiton of the surrounding structures of thord molar teeth was assessed (periodontally affected or not).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No